CLINICAL TRIAL: NCT04713670
Title: Comparison of Vonoprazan-based Versus Lansoprazole-based Triple Therapy, High Dose Dual Therapy, Bismuth and Non-bismuth Quadruple Therapy in the First-line Treatment of Helicobacter Pylori Infection - a Multicenter, Open Labelled, Randomized Pilot Trial
Brief Title: Comparison of Vonoprazan-based Versus Lansoprazole-based Triple Therapy, High Dose Dual Therapy, Bismuth and Non-bismuth Quadruple Therapy in the First-line Treatment of Helicobacter Pylori Infection
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202004063MINA
Record Dates: First submitted 2021-01-10; First posted 2021-01-19 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: H. Pylori Infection
Keywords: H.pylori; vonoprazan; lansoprazole; triple therapy; high dose dual therapy; bismuth quadruple
MeSH Terms: interventions — Fumigant 93; Protons

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- (A) T-V14 (Experimental)
  Interventions: Drug: (A) T-V14
- (B) T-V7 (Experimental)
  Interventions: Drug: (B) T-V7
- (C) D-V14 (Experimental)
  Interventions: Drug: (C) D-V14
- (D) HD-V14 (Experimental)
  Interventions: Drug: (D) HD-V14
- (E) BQ-V14 (Experimental)
  Interventions: Drug: (E) BQ-V14
- (F) RH-V14 (Experimental)
  Interventions: Drug: (F) RH-V14
- (G) BQ-L14 (Experimental)
  Interventions: Drug: (G) BQ-L14
- (H) T-L14 (Experimental)
  Interventions: Drug: (H) T-L14

INTERVENTIONS:
Drug: (A) T-V14 — vonoprazan(vocinti)-based triple therapy for 14 days (T-V14)
  Arms: (A) T-V14
Drug: (B) T-V7 — vonoprazan(vocinti)-based triple therapy for 7 days (T-V7)
  Arms: (B) T-V7
Drug: (C) D-V14 — vonoprazan(vocinti)-based dual therapy for 14 days (D-V14)
  Arms: (C) D-V14
Drug: (D) HD-V14 — vonoprazan(vocinti)-based high dose dual therapy for 14 days (HD-V14)
  Arms: (D) HD-V14
Drug: (E) BQ-V14 — vonoprazan(vocinti)-based bismuth quadruple therapy for 14 days (BQ-V14)
  Arms: (E) BQ-V14
Drug: (F) RH-V14 — vonoprazan(vocinti)-based reverse hybrid therapy for 14 days (RH-V14)
  Arms: (F) RH-V14
Drug: (G) BQ-L14 — lansoprazole(takepron)-based bismuth quadruple therapy for 14 days (BQ-L14)
  Arms: (G) BQ-L14
Drug: (H) T-L14 — lansoprazole(takepron)-based triple therapy for 14 days (T-L14)
  Arms: (H) T-L14

SUMMARY:
Background: Bismuth quadruple therapy is currently the recommended first-line regimen for Helicobacter pylori (H. pylori) infection in regions with high clarithromycin resistance. Recent randomized trials showed that 7-day vonoprazan-based triple therapy is superior to 7-day lansoprazole-based triple therapy in Japanese. A recent trial further showed that 7-day vonoprazan-based high dose amoxicillin dual therapy was non-inferior to 7-day vonoprazan-based triple therapy in Japanese. However, whether vonoprazan based dual, triple, and quadruple therapies are superior or non-inferior to lansoprazole based triple or quadruple therapy remains unknown.

Objective: The investigators aimed to compare the efficacy and safety of 14-day vonoprazan-based dual therapy, triple therapy, bismuth quadruple therapy, reverse hybrid therapy, and lansoprazole-based bismuth quadruple therapy and triple therapy in the first-line treatment of H. pylori infection in this pilot study.

Methods: Using a block randomization with a block size of 16 in a 1:1 ratio, 1200 eligible adult subjects aged 20 years or greater with at least two positive tests for H. pylori infection will be randomized to receive one of the following regimens: (A) vonoprazan-based triple therapy for 14 days (T-V14): vonoprazan 20mg twice daily, clarithromycin-XL 500mg twice daily, amoxicillin 1000mg twice daily for 14 days ; or (B) vonoprazan-based triple therapy for 7 days (T-V7): vonoprazan 20mg twice daily, clarithromycin-XL 500mg twice daily, amoxicillin 1000mg twice daily for 7 days ; or (C): vonoprazan-based dual therapy for 14 days (D-V14): vonoprazan 20mg twice daily, amoxicillin 750mg every 8 hour for 14 days; (D): vonoprazan-based high dose dual therapy for 14 days (HD-V14): vonoprazan 20mg twice daily, amoxicillin 750mg four times a day for 14 days; or (E) vonoprazan-based bismuth quadruple therapy for 14 days (BQ-V14) vonoprazan 20mg twice daily, bismuth tripotassium dicitrate 300 mg three times a day, tetracycline 500mg three times a day, and metronidazole 500mg three times a day for 14 days; or (F) vonoprazan-based reverse hybrid therapy for 14 days (RH-V14): vonoprazan 20mg twice daily, and amoxicillin 1000mg twice daily for 14 days, plus clarithromycin-XL 500mg twice daily and metronidazole 500mg twice daily for the first 7 days ; or (G) lansoprazole-based bismuth quadruple therapy for 14 days (BQ-L14) lansoprazole 30mg twice daily, bismuth tripotassium dicitrate 300 mg three times a day, tetracycline 500mg three times a day, and metronidazole 500mg three times a day for 14 days; or (H) lansoprazole-based triple therapy for 14 days (T-L14): lansoprazole 30mg twice daily, clarithromycin-XL 500mg twice daily, amoxicillin 1000mg twice daily for 14 days. Subjects who fail after first-line therapy will be randomized to receive either vonoprazan-based levofloxacin triple therapy (LT-V14) containing vonoprazan 20mg twice daily, levofloxacin 250mg twice daily, and amoxicillin 1000mg twice daily for 14 days or vonoprazan-based levofloxacin reverse hybrid therapy (LRH-V14) containing vonoprazan 20mg twice daily, and amoxicillin 1000mg twice daily for 14 days, plus levofloxacin 250mg twice daily and metronidazole 500mg twice daily for the first 7 days. The minimum inhibitory concentrations will be determined by agar dilution test. 23S ribosomal RNA and gyrase A mutations will be determined by PCR methods followed by direct sequencing in a subgroup of patients. The TWB2.0 SNP array will be used for genotyping of genome wide single nucleotide polymorphism.

Outcome analysis: The primary outcome is the eradication rate in the first-line treatment. The secondary outcomes are the compliance, frequency of adverse events, the overall eradication rate after two treatments.

DETAILED DESCRIPTION:
Background: Bismuth quadruple therapy is currently the recommended first-line regimen for Helicobacter pylori (H. pylori) infection in regions with high clarithromycin resistance. Recent randomized trials showed that 7-day vonoprazan-based triple therapy is superior to 7-day lansoprazole-based triple therapy in Japanese. A recent trial further showed that 7-day vonoprazan-based high dose amoxicillin dual therapy was non-inferior to 7-day vonoprazan-based triple therapy in Japanese. However, whether vonoprazan based dual, triple, and quadruple therapies are superior or non-inferior to lansoprazole based triple or quadruple therapy remains unknown.

Objective: The investigators aimed to compare the efficacy and safety of 14-day vonoprazan-based dual therapy, triple therapy, bismuth quadruple therapy, reverse hybrid therapy, and lansoprazole-based bismuth quadruple therapy and triple therapy in the first-line treatment of H. pylori infection in this pilot study. The long-term changes in gut microbiota, antibiotic resistance, trimethylamine-N-oxide (TMAO) levels, and metabolic parameters after eradication therapies will also be investigated.

Methods: Using a block randomization with a block size of 16 in a 1:1 ratio, 1200 eligible adult subjects aged 20 years or greater with at least two positive tests for H. pylori infection will be randomized to receive one of the following regimens: (A) vonoprazan-based triple therapy for 14 days (T-V14): vonoprazan 20mg twice daily, clarithromycin-XL 500mg twice daily, amoxicillin 1000mg twice daily for 14 days ; or (B) vonoprazan-based triple therapy for 7 days (T-V7): vonoprazan 20mg twice daily, clarithromycin-XL 500mg twice daily, amoxicillin 1000mg twice daily for 7 days ; or (C): vonoprazan-based dual therapy for 14 days (D-V14): vonoprazan 20mg twice daily, amoxicillin 750mg every 8 hour for 14 days; (D): vonoprazan-based high dose dual therapy for 14 days (HD-V14): vonoprazan 20mg twice daily, amoxicillin 750mg four times a day for 14 days; or (E) vonoprazan-based bismuth quadruple therapy for 14 days (BQ-V14) vonoprazan 20mg twice daily, bismuth tripotassium dicitrate 300 mg three times a day, tetracycline 500mg three times a day, and metronidazole 500mg three times a day for 14 days; or (F) vonoprazan-based reverse hybrid therapy for 14 days (RH-V14): vonoprazan 20mg twice daily, and amoxicillin 1000mg twice daily for 14 days, plus clarithromycin-XL 500mg twice daily and metronidazole 500mg twice daily for the first 7 days ; or (G) lansoprazole-based bismuth quadruple therapy for 14 days (BQ-L14) lansoprazole 30mg twice daily, bismuth tripotassium dicitrate 300 mg three times a day, tetracycline 500mg three times a day, and metronidazole 500mg three times a day for 14 days; or (H) lansoprazole-based triple therapy for 14 days (T-L14): lansoprazole 30mg twice daily, clarithromycin-XL 500mg twice daily, amoxicillin 1000mg twice daily for 14 days. Subjects who fail after first-line therapy will be randomized to receive either vonoprazan-based levofloxacin triple therapy (LT-V14) containing vonoprazan 20mg twice daily, levofloxacin 250mg twice daily, and amoxicillin 1000mg twice daily for 14 days or vonoprazan-based levofloxacin reverse hybrid therapy (LRH-V14) containing vonoprazan 20mg twice daily, and amoxicillin 1000mg twice daily for 14 days, plus levofloxacin 250mg twice daily and metronidazole 500mg twice daily for the first 7 days. The minimum inhibitory concentrations will be determined by agar dilution test. 23S ribosomal RNA and gyrase A mutations will be determined by PCR methods followed by direct sequencing in a subgroup of patients. The TWB2.0 SNP array will be used for genotyping of genome wide single nucleotide polymorphism. Fecal and oral samples will be collected for 16S and shot-gun sequencing at baseline, week 2, week 8, year 1, and year 2. Metabolic parameters will be measured at baseline, week 8, year 1, and year 2. Modified carnitine challenge test (mCCT) will be done to assess the production of urine TMAO at baseline, week 2, week 8, year 1, and year 2 in a subgroup of study subjects.

Outcome analysis: The primary outcome is the eradication rate in the first-line treatment. The secondary outcomes are the compliance, frequency of adverse events, the overall eradication rate after two treatments. The long-term outcomes are the cumulative eradication rate, the changes of gut microbiota, antibiotic resistance, TMAO production, and metabolic parameters at year 1 and year 2.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with naive H. pylori infection
2. Subjects with over 20 years old

Exclusion Criteria:

1. Younger than 20 years old
2. Ever received H. eradication therapy
3. ever received total or subtotal gastrectomy in the past
4. Severe chronic disease, such as end stage renal disease, liver cirrhosis, incurable malignant tumors
5. Women who are pregnant or breastfeeding
6. Those who are not suitable to receive study drugs: such as a history of allergies to study drugs or serious side effects, etc.
7. Patients with chronic hepatitis (AST or ALT >40 IU/L)
8. Subjects who cannot sign informed consent by themselves

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the eradication rate in the first-line treatment. | Up to 8-12 weeks
  At least 6 weeks after the end of treatment, the carbon 13-breath test will be used to evaluate whether the eradication is successful. The eradication rate in each group will be presented as "%"

SECONDARY OUTCOMES:
The secondary outcomes are the compliance and frequency of adverse events. | Up to 8-12 weeks
  After eradication treatment, participants will go back to the outpatients clinics to evaluate whether they take all of or > 80% drugs. The investigators will also record any side effect associated with treatment, such as skin rash, dizziness, headache, taste distortion, and etc. The severity grading include "none", "mild", "moderate", "severe" and "life-threatening".

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Ming Liou, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan